CLINICAL TRIAL: NCT04934553
Title: Amplification of Positivity for Alcohol Use Disorder (AMP-A): Feasibility and Pilot Study
Brief Title: Amplification of Positivity for Alcohol Use Disorder Co-Occurring With Anxiety or Depression
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Limited funding
Sponsor: Charles Taylor (Other)
Collaborators: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Sponsor-Investigator, Charles Taylor, Assoc Adjt Prof, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 210136
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Alcoholism; Alcohol Drinking; Drinking Behavior; Alcohol-Related Disorders; Substance-Related Disorders; Mental Disorder; Anxiety; Depression
MeSH Terms: conditions — Alcoholism; Alcohol Drinking; Drinking Behavior; Alcohol-Related Disorders; Substance-Related Disorders; Mental Disorders; Anxiety Disorders; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amplification of Positivity for Alcohol Use Disorders (AMP-A; 12 sessions) (Experimental)
  Interventions: Behavioral: Amplification of Positivity Training
- Cognitive-behavioral Therapy (CBT; 12 sessions) (Active Comparator)
  Interventions: Behavioral: Cognitive-behavioral Therapy

INTERVENTIONS:
Behavioral: Amplification of Positivity Training — 12 90-minute, clinician-administered treatment sessions focused on presenting rationale and instructions for completing positive activity exercises (e.g., gratitude, acts of kindness) designed to increase positive emotions, cognitions, and behaviors.
  Arms: Amplification of Positivity for Alcohol Use Disorders (AMP-A; 12 sessions)
Behavioral: Cognitive-behavioral Therapy — 12 90-minute, clinician-administered treatment sessions focused on strategies to alter cognitions and behavior related to alcohol use.
  Arms: Cognitive-behavioral Therapy (CBT; 12 sessions)

SUMMARY:
The purpose of this study is to examine the feasibility of a protocol in which individuals with comorbid depression or anxiety disorders and alcohol use disorder will be randomized to complete Amplification of Positivity for Alcohol Use Disorder (AMP-A)- a psychological treatment focused on increasing positive thoughts, emotions, and behaviors- or a traditional cognitive-behavioral therapy (CBT) intervention. Assessed outcomes will include participant acceptability and completion rates, participant compliance with the intervention, positive and negative affect, substance use- and depression and anxiety-related symptom severity, and functional disability.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 55 years old.
* Meet diagnostic criteria for alcohol use disorder according to the DSM-5
* Significant depression or anxiety symptoms as indexed by scoring Patient Health Questionnaire (PHQ-9) ≥ 10 and/or Overall Anxiety Severity and Impairment Scale (OASIS) ≥ 8.
* Able to provide written informed consent.
* Have sufficient proficiency in the English language to understand and complete interviews, questionnaires, and all other study procedures.
* Completion of at least an 8th grade education, to help facilitate ability to engage in the written materials included in the treatments.

Exclusion Criteria:

* Unwillingness or inability to complete any of the major aspects of the study protocol, including self-report or behavioral assessment. However, failing to complete some individual aspects of these assessment sessions will be acceptable (i.e., being unwilling to answer individual items on some questionnaires or being unwilling to complete a behavioral task).
* Non-correctable vision or hearing problems.
* No telephone or easy access to telephone.
* Diagnosis of Schizophrenia spectrum, other psychotic disorders, or bipolar I disorder.
* Active suicidal ideation with plan and intent to attempt suicide within the next month.
* Has a history of unstable liver or renal insufficiency; glaucoma; significant and unstable cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, or metabolic disturbance; or any other condition that, in the opinion of the investigator, would make participation not be in the best interest (e.g., compromise the well-being) of the subject or that could prevent, limit, or confound the protocol-specified assessments.
* A positive test for alcohol (breath test) at the time of baseline assessments. Participants will be asked to refrain from using alcohol within 24 hours prior to assessment sessions and to refrain from using marijuana within 48 hours of assessment sessions.
* Initiation of a new psychotropic medication (e.g., SSRIs) or change in the dose or prescription of a medication within the 6 weeks prior to enrolling in the study.
* Concurrent engagement in psychosocial treatments that specifically target alcohol use disorder or mood/anxiety symptoms and began within 12 weeks of baseline assessments. Individuals concurrently receiving psychosocial treatments for other symptoms, or that are not specifically targeting symptoms (e.g., ongoing support groups) will not be excluded as long as the dose of treatment (i.e., frequency of sessions) has not changed significantly within 6 weeks prior to enrolling in the study.
* Moderate to severe traumatic brain injury (>30 min. loss of consciousness or >24 hours posttraumatic amnesia) or other neurocognitive disorder with evidence of neurological deficits, neurological disorders, or severe or unstable medical conditions that might be compromised by participation in the study (to be determined by primary care provider).
* Severity of alcohol use disorder requiring more intensive treatment (i.e., intensive outpatient or residential), as determined by baseline assessments conducted by clinicians.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Adherence and Acceptability Scale (AAS) | Post intervention (approximately 2 weeks after completing intervention)
  The AAS assesses the acceptability and tolerability of the intervention. Scores may range from 10 to 70, with higher scores indicating greater acceptability of treatment and greater anticipated ability to adhere to it.
Distress/Endorsement Validation Scale (DEVS) | Post intervention (approximately 2 weeks after completing intervention)
  The DEVS measure assesses two factors, distress (7 items) and endorsement (3 items). The distress subscale score ranges from 7 to 63, with higher scores indicating more distress experienced during the intervention. The endorsement subscale ranges from 3 to 27, with higher scores indicating greater endorsement of the intervention.
Completion rate | Post intervention (approximately 2 weeks after completing intervention)
  Completion rate assessed as whether or not the participant completes all 12 sessions of intervention

SECONDARY OUTCOMES:
Change from baseline in well-being as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Positive Affect and Well-being Scale | Baseline, Primary Endpoint: Post-treatment (i.e., within two weeks of completing the intervention), Secondary Endpoints: Three month follow-up (i.e., 12-15 weeks after completing the intervention)
  The PROMIS Positive Affect and Well-being Scale assesses positive or rewarding affective experiences over the past 7 days. The score is presented as a T score with a mean of 50 and standard deviation of 10, with higher scores indicating greater positive affect and well-being.
Change from baseline in alcohol craving as measured by the Alcohol Craving Questionnaire (ACQ) | Baseline, Primary Endpoint: Post-treatment (i.e., within two weeks of completing the intervention), Secondary Endpoints: Three month follow-up (i.e., 12-15 weeks after completing the intervention)
  The ACQ assesses four dimensions of alcohol craving. A total score ranges from 1-12, with higher scores indicating higher levels of alcohol craving.
Change from baseline in positive affect as measured by Positive and Negative Affect Schedule | Baseline, Primary Endpoint: Post-treatment (i.e., within two weeks of completing the intervention), Secondary Endpoints: Three month follow-up (i.e., 12-15 weeks after completing the intervention)
  The Positive and Negative Affect Schedule (PANAS) measures positive affect. Items are answered on a 5 point scale, 1 (Very slightly or not at all) to 5 (Extremely). The positive affect scale ranges from 10-50 and higher scores indicate greater levels of positive affect.
Change from baseline in anxiety as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Scale | Baseline, Primary Endpoint: Post-treatment (i.e., within two weeks of completing the intervention), Secondary Endpoints: Three month follow-up (i.e., 12-15 weeks after completing the intervention)
  The PROMIS Anxiety scale assesses symptoms of anxiety over the past 7 days. The score is presented as a T score with a mean of 50 and standard deviation of 10, with higher scores indicating greater symptoms of anxiety.
Change from baseline in depression as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Scale | Baseline, Primary Endpoint: Post-treatment (i.e., within two weeks of completing the intervention), Secondary Endpoints: Three month follow-up (i.e., 12-15 weeks after completing the intervention)
  The PROMIS Depression scale assesses symptoms of depression over the past 7 days. The score is presented as a T score with a mean of 50 and standard deviation of 10, with higher scores indicating greater symptoms of depression.
Change from baseline in level of functional disability as measured by the Sheehan Disability Scale (SDS) | Baseline, Primary Endpoint: Post-treatment (i.e., within two weeks of completing the intervention), Secondary Endpoints: Three month follow-up (i.e., 12-15 weeks after completing the intervention)
  The SDS assesses level of functional disability. Total score ranges from 0-30, with higher scores indicating greater impairment.
Change from baseline in alcohol use | Baseline, Primary Endpoint: Post-treatment (i.e., within two weeks of completing the intervention), Secondary Endpoints: Three month follow-up (i.e., 12-15 weeks after completing the intervention)
  As measured by self-reported drinks per day
Change from baseline in pleasure experience as measured by the Snaith-Hamilton Please Scale (SHAPS) | Baseline, Primary Endpoint: Post-treatment (i.e., within two weeks of completing the intervention), Secondary Endpoints: Three month follow-up (i.e., 12-15 weeks after completing the intervention)
  The SHAPS assesses the ability to experience pleasure. Total scores range from 0 to 14, with a higher score indicating higher levels of anhedonia.

CONTACTS AND LOCATIONS:
Overall Officials: Charles T Taylor, PhD, Principal Investigator — Altman Clinical and Translational Research Institute; Robin Aupperle, PhD, Principal Investigator — Laureate Institute for Brain Research
Locations (2):
- United States (2):
  - Altman Clinical and Translational Research Institute, La Jolla, California
  - Laureate Institute for Brain Research, Tulsa, Oklahoma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taylor CT, Lyubomirsky S, Stein MB. Upregulating the positive affect system in anxiety and depression: Outcomes of a positive activity intervention. Depress Anxiety. 2017 Mar;34(3):267-280. doi: 10.1002/da.22593. Epub 2017 Jan 6. PMID 28060463